CLINICAL TRIAL: NCT06809283
Title: Observational Prospective Post Market Clinical Follow-up (PMCF) Study to Confirm the Performance and Safety of the Chattanooga Intelect® Devices in Real World Use
Brief Title: Observational Prospective PMCF Study to Confirm Performance and Safety of Intelect® Devices in Real World
Acronym: INTELECT
Status: Recruiting | Type: Observational
Sponsor: DJO UK Ltd (Industry)
Collaborators: Donawa Lifescience Consulting SRL (Unknown)
Responsible Party: Sponsor
Other Study IDs: ENOVIS-S-INP-0004
Record Dates: First submitted 2025-01-27; First posted 2025-02-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Musculoskeletal Disorders; Skeletal Disorder; Muscle Disorder
Keywords: TENS; NMES; Ultrasound; Pain; ROM
MeSH Terms: conditions — Musculoskeletal Diseases; Muscular Diseases; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TENS/US group: Patient affected by acute or chronic musculoskeletal pain or affected by post-operative pain that will be treated with TENS alone, US alone or TENS + US according to the current standard clinical practice at site.
  Data from patients in this group will be used to determine the primary study objective, some of the exploratory objectives and the safety objectives.
- NMES group: Patients affected by skeletal muscle deficit disorders who benefit form muscle re-education and/or maintaining/increasing the range of motion will be treated with NMES alone or NMES + US according to the current standard clinical practice at site.
  Data from patients in this group will be used to determine the secondary study objective, some of the exploratory objectives and the safety objectives

SUMMARY:
DJO UK Ltd (ENOVIS) is conducting this study to confirm the performance and safety of the Chattanooga Intelect® devices in real world use. This study will record post market clinical data on the use of a number of MDR-CE marked devices that are part of the Chattanooga Intelect® device family to ensure the continued acceptability of the benefit-risk ratio, and to identify possible systematic misuse or off-label use of the devices (Intelect® Mobile 2 Combo, Intelect® Mobile 2 Ultrasound, Intelect® Mobile 2 Electrotherapy (Stim), Intelect® Transport 2 Combo and Intelect® Transport 2 Ultrasound).

DETAILED DESCRIPTION:
This clinical investigation is a post-market, real word, international, multi center, prospective, observational study to confirm the safety and performance of the Chattanooga Intelect® when used in accordance with their approved intended use, to comply with Medical Device Regulation (EU) 2017/745 (MDR) Article 61 and Part B of Annex XI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with musculoskeletal and skeletal muscle deficit disorders assigned to be treated with any of the Intelect® devices according to the current clinical practice at the selected sites and based on the opinion of the Investigator.
2. Patient male or female with age ≥18 years old.
3. Patient able to provide written informed consent. For France only: To be affiliated to the social security system or to be beneficiary of such system

Exclusion Criteria:

1. Patients participating in another clinical study or who have completed a clinical study less than 30 days prior to enrollment.
2. Patients who for any reason e.g. significant co-morbidities or other reasons, are considered by the Investigator unsuitable for study participation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with musculoskeletal and skeletal muscle deficit disorders planned to be treated with any of the Intelect® devices who spontaneously went to any of the selected sites for receiving a treatment. For the purpose of determining the type of performance data to be collected, patients will be assigned to two groups: TENS/US group or NMES group based on the treatment they receive during their first session.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | from treatment start to treatment end (about 6 weeks)
  Pain reduction measured with Visual Analog Scale (VAS) (in a scale 0-100 mm, where 0 is no pain and 100 is the worst possible pain) at end of treatment compared to pre-treatment (baseline) VAS in the TENS/US group

SECONDARY OUTCOMES:
Muscle reeducation | from treatment start to treatment end (about 6 weeks)
  Improvement in muscle re-education demonstrated by score on a digital dynamometer at the end of treatment compared to baseline in the NMES group
Range of motion (ROM) improvement | from treatment start to treatment end (about 6 weeks)
  Maintenance or increasing of the ROM demonstrated by a goniometer the end of treatment compared to baseline in the NMES group
Clinical status improvement | end of study (about 12 weeks)
  Improvement in patient clinical status using the Global Clinical Assessment of improvement questionnaire at the end of the treatment in the NMES group
Safety - adverse event rate | through study completion, an average of 15 weeks
  Proportion of patient experiencing an adverse event associated with device use

OTHER OUTCOMES:
Waveforms assessment | through study completion, an average of 15 weeks
  Assess the performance and safety of the different waveforms used in the TENS and NMES modalities
Electrodes assessment | through study completion, an average of 15 weeks
  Assess the performance and safety of various types of electrodes used with the Intelect® devices for TENS or NEMS modalities
Misuse or off-label use identification | end of treatment (about 6 weeks)
  Identify misuse or off-label use of the Intelect® devices

CONTACTS AND LOCATIONS:
Locations (4):
- Attal Cabinet, Serris, France
- Italy (2):
  - Casertafisio, Caserta
  - Rachis Center, Roma
- Dr Chad Woods Physiotherapy, Peebles, United Kingdom